CLINICAL TRIAL: NCT04131543
Title: "Phase II Study to Evaluate the Activity and Safety of Cabozantinib in Pretreated, Advanced RET-rearranged Non-small Cell Lung Cancer Patients: CRETA Trial"
Brief Title: Phase II Study With Cabozantinib in Patients With RET Positive NSCLC
Acronym: CRETA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Collaborators: AOU S.Orsola Malpighi-Unit of Oncologic Molecular and Transplantations Pathology (Unknown); Bioikos Ambiente Srl (Other); Ipsen (Industry); Mipharm SpA (Unknown)
Responsible Party: Principal Investigator, Andrea Ardizzoni, Professor/MD, University of Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRETA
Record Dates: First submitted 2019-09-26; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: Single-arm, ope label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): Cabozantinib will be administered orally at a (starting) dose of 60 mg once daily. The drug is taken continuously over a period of 28 days (4 weeks), which constitutes one treatment cycle. In all subjects, dose reductions and delays to manage toxicity. Cabozantinib should be taken in fasting condition with no food for at least 2 hours before and 1 hour after taking the tablets. A high fat meal significantly increased the median tmax to 6 hours from 4 hours (fasted). The treatment will be continued until disease progression, intolerable toxicity, patient refusal or Investigator's decision or any criterion for withdrawal from the trial or trial drug is fulfilled.
  Interventions: Drug: Cabozantinib 20 MG; Drug: Cabozantinib 40 MG; Drug: Cabozantinib 60 MG

INTERVENTIONS:
Drug: Cabozantinib 20 MG — Cabozantinib will be administered orally at a (starting) dose of 60 mg once daily. The drug is taken continuously over a period of 28 days (4 weeks), which constitutes one treatment cycle. In all subjects, dose reductions (40mg 20mg) and delays to manage toxicity.
  Other Names: CABOMETYX
Drug: Cabozantinib 40 MG — Cabozantinib will be administered orally at a (starting) dose of 60 mg once daily. The drug is taken continuously over a period of 28 days (4 weeks), which constitutes one treatment cycle. In all subjects, dose reductions (40mg 20mg) and delays to manage toxicity.
  Other Names: CABOMETYX
Drug: Cabozantinib 60 MG — Cabozantinib will be administered orally at a (starting) dose of 60 mg once daily. The drug is taken continuously over a period of 28 days (4 weeks), which constitutes one treatment cycle. In all subjects, dose reductions and delays to manage toxicity. Cabozantinib should be taken in fasting condition with no food for at least 2 hours before and 1 hour after taking the tablets. A high fat meal significantly increased the median tmax to 6 hours from 4 hours (fasted). The treatment will be continued until disease progression, intolerable toxicity, patient refusal or Investigator's decision or any criterion for withdrawal from the trial or trial drug is fulfilled.
  Other Names: CABOMETYX

SUMMARY:
This study is aimed to explore the antitumor activity, safety and efficacy profile of cabozantinib in pretreated, advanced RET-rearranged non-small cell lung cancer patients

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced, relapsed or metastatic non-small cell lung cancer - stage IIIB/IV according to 7th International Association for the Study of Lung Cancer (IASLC) classification
2. Ability to understand and willingness to sign informed consent prior to initiation of any study procedures.
3. Pathologically (histology or cytology) confirmed diagnosis of non- small cell lung carcinoma.
4. RET gene rearrangement by local laboratory analysis with an approved standard method (FISH or Next Generation Sequencing Panel). An archival tumor sample must be available for central laboratory confirmation.
5. Male or female and = 18 years of age
6. Life expectancy = 12 weeks
7. Have progressed after or during at least one standard anticancer treatment
8. Have measurable disease as per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1); clear radiological evidence of disease progression after first-line therapy must be documented; no previous radiotherapy on the only site of measurable or evaluable disease, unless that site had subsequent evidence of progression
9. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 1
10. Subjects must have adequate organ function including the following:

    * Absolute neutrophil count > 1.5 x 10^9/L
    * Platelet count > 100 x 10^9/L
    * Haemoglobin > 90 g/L
    * ALT < 2.5 times the upper limit of normal (ULN)
    * AST < 2.5 times ULN
    * Total bilirubin <1.5 times ULN
    * Creatinine <1.5 times ULN concurrent with creatinine clearance > 50 ml/min (measured or calculated by Cockcroft and Gault equation, confirmation of creatinine clearance is only required when creatinine is > 1.5 times ULN)
    * Lipase < 2.0 times the upper limit of normal (ULN)
11. Stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections, or major surgery within 4 weeks before registration, and otherwise noted in other inclusion/exclusion criteria
12. Recovered (i.e., = Grade 1 toxicity) from effects of prior anticancer therapy, except alopecia
13. No radiologic or clinical evidence of acute or chronic pancreatitis
14. For Females: must be postmenopausal (defined as amenhorrea = 12 consecutive months) before the screening visit, or are surgically sterile. If they are of childbearing potential, a negative serum pregnancy test obtained within 3 days before starting study treatment has to be documented; furthermore, patients must agree to adopt 2 effective methods of contraception, at the same time, from the time of signing the informed consent form (ICF) through 4 months after the last dose of study drug.
15. For Males: even if surgically sterilized (i.e. post-vasectomy status) agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug.
16. Ability to comply with protocol requirement.

Exclusion criteria:

1. Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before randomization. Systemic treatment with radionuclides within 6 weeks before randomization. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
2. Previous treatment with cabozantinib.
3. Gastrointestinal disorders likely to interfere with absorption of the study drug.
4. Subjects with gastrointestinal disorders associated with a high risk of perforation of fistula formation.
5. Subjects with active peptic ulcer or with a history of clinically ¿significant GI bleeding within 6 months before the first dose of study treatment.
6. Patients requiring full-dose anticoagulation therapy any time prior to enrollment.
7. Current use of aspirin, clopidogrel, ticlopidine.
8. Patients with tumors invading major pulmonary vessels and/or with cavitating pulmonary lesions.
9. Major surgery within the last four weeks. Complete wound healing from major surgery must have occurred 1 month before randomization and from minor surgery at least 10 days before randomization. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
10. Subjects with clinical or radiological signs of pulmonary hemorrhage within 3 months before the first dose of study treatment.
11. Symptomatic CNS or leptomeningeal lesions, not previously treated with radiotherapy.

    Untreated central nervous system (CNS) or leptomeningeal metastases are allowed if asymptomatic. Patients with symptomatic CNS or leptomeningeal lesions will be allowed to participate in this study if previously treated with radiotherapy and on stable dose of corticosteroids and/or anticonvulsants for > 10 days or not requiring such medication.

    Radiotherapy must have been completed a minimum of 4 weeks prior to registration, and patients must have recovered from AEs related to radiotherapy to < grade 1 (except alopecia).
12. History of congenital platelet function defect.
13. Patient unable to swallow tablets
14. Corrected QT interval greater than 500 ms (Fridericia formula)
15. Clinically significant, uncontrolled heart diseases:

    * Unstable angina within 6 months prior to screening
    * Myocardial infarction within 6 months prior to screening
    * History of documented congestive heart failure
    * Uncontrolled hypertension defined by a Systolic Blood Pressure , with or without antihypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening
    * Ventricular arrhythmias, Supraventricular and nodal arrhythmias not controlled with medication
    * Congenital history of QT syndrome.
16. Diagnosed with or treated for another malignancy within 3 years before the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type may be enrolled in the study if they have undergone complete resection and no evidence of active disease is present.
17. Any type of systemic anticancer agent within 3 weeks of first dose of study treatment, or within 5 half- lives of the agent whichever is shorter (subjects on LHRH or GnRH agonists may be maintained on these agents)
18. Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
19. Rare hereditary problems of

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-08-07 (Actual); Primary Completion 2020-08-07 (Estimated); Study Completion 2022-08-07 (Estimated)

PRIMARY OUTCOMES:
Response Rate (RR) | From the start of treatment ( Baseline) to the progression of Disease (PD) or trial discontinuation whichever occurs first, assessed up to 24 months
  Exact binomial method will be used to estimate the response rate (CR+PR) and its 95% confidence interval.Proportion of patients presenting Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) based on the Investigator's assessment according to standard RECIST criteria v1.1. Patients with no tumor assessment after baseline will be classified as non-responders.

SECONDARY OUTCOMES:
Toxicity (frequency of adverse events) | From the start of treatment ( Baseline) to the progression of Disease (PD) or trial discontinuation whichever occurs first, assessed up to 24 months
  the assessment of safety will be based mainly on the frequency of adverse events; toxicity will be measured according to NCI Common Toxicity Criteria Adverse Event (CTCAE), version 4.03.
Progression-Free Survival (PFS) | From the start of treatment ( Baseline) to the progression of Disease (PD) or trial discontinuation whichever occurs first, assessed up to 24 months
  PFS will be calculated from the first treatment intake to the date of progressive disease, or death.
Overall survival (OS) | From the start of treatment ( Baseline) to the progression of Disease (PD) or trial discontinuation whichever occurs first, assessed up to 24 months
  OS will be calculated from the first treatment intake to death from any cause.
Duration of response (DOR | From the start of treatment ( Baseline) to the progression of Disease (PD) or trial discontinuation whichever occurs first, assessed up to 24 months
  DOR will be calculated from the first treatment intake to the date of disease progression or death.
Disease Control Rate(DCR) | From the start of treatment ( Baseline) to the progression of Disease (PD) or trial discontinuation whichever occurs first, assessed up to 24 months
  DCR will be measured as the sum of complete and partial responses + stable disease.

OTHER OUTCOMES:
RET aberration | On the start of treatment (Baseline) and through study completion, an average of 1 year
  Detection of RET aberration on DNA extracted from circulating tumor cells (CTCs) isolated in blood at baseline (optional)
RET-rearrangment on tumor tissue | At the start of treatment (baseline)
  Archival tumor tissue (FFPE tumor block or 7-10 unstained slides) will be assessed for determination of RET-rearrangment on tumor cells by using A FISH evaluation of the translocation will be performed using a break-apart probe for the 10p11 locus.

CONTACTS AND LOCATIONS:
Locations (11):
- Italy (11):
  - OU di Oncologia Medica- Azienda ospedaliero-Universitaria S. Orsola Malpighi, Bologna
  - U.O di Oncologia Medica Policlinico V.Emanuele-G.Rodolico, Catania
  - Oncologia Medica 2 -Policlinico San Martino, Genova
  - S.S. di Oncologia Medica toraco-polmonare - Fondazione IRCCS - Istituto Nazionale Tumori, Milan
  - U.O.C Pneumologia ad Indirizzo Oncologico -AORN Ospedali dei Colli Monaldi-Cotugno-CTO, Napoli
  - UOC di Oncologia Medica 2 - IOV Istituto Oncologico Veneto, Padua
  - UOC di Oncologia Medica- Azienda Ospidaliero Universitaria di Parma, Parma
  - US di Oncologia Medica - A.O. di Perugia, Perugia
  - UO Pneumologia - A.O.U Pisana, Pisa
  - S.C. di Oncologia Medica - IFO - Istituto Regina Elena, Roma
  - UOC di Oncologia Medica - Azienda Sanitaria Universitaria Integrata di Udine, Udine

REFERENCES:
- [Result] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Result] Masters GA, Temin S, Azzoli CG, Giaccone G, Baker S Jr, Brahmer JR, Ellis PM, Gajra A, Rackear N, Schiller JH, Smith TJ, Strawn JR, Trent D, Johnson DH; American Society of Clinical Oncology Clinical Practice. Systemic Therapy for Stage IV Non-Small-Cell Lung Cancer: American Society of Clinical Oncology Clinical Practice Guideline Update. J Clin Oncol. 2015 Oct 20;33(30):3488-515. doi: 10.1200/JCO.2015.62.1342. Epub 2015 Aug 31. PMID 26324367
- [Result] Zbuk KM, Eng C. Cancer phenomics: RET and PTEN as illustrative models. Nat Rev Cancer. 2007 Jan;7(1):35-45. doi: 10.1038/nrc2037. Epub 2006 Dec 14. PMID 17167516
- [Result] Grieco M, Santoro M, Berlingieri MT, Melillo RM, Donghi R, Bongarzone I, Pierotti MA, Della Porta G, Fusco A, Vecchio G. PTC is a novel rearranged form of the ret proto-oncogene and is frequently detected in vivo in human thyroid papillary carcinomas. Cell. 1990 Feb 23;60(4):557-63. doi: 10.1016/0092-8674(90)90659-3. PMID 2406025
- [Result] Bongarzone I, Vigneri P, Mariani L, Collini P, Pilotti S, Pierotti MA. RET/NTRK1 rearrangements in thyroid gland tumors of the papillary carcinoma family: correlation with clinicopathological features. Clin Cancer Res. 1998 Jan;4(1):223-8. PMID 9516975
- [Result] Wang R, Hu H, Pan Y, Li Y, Ye T, Li C, Luo X, Wang L, Li H, Zhang Y, Li F, Lu Y, Lu Q, Xu J, Garfield D, Shen L, Ji H, Pao W, Sun Y, Chen H. RET fusions define a unique molecular and clinicopathologic subtype of non-small-cell lung cancer. J Clin Oncol. 2012 Dec 10;30(35):4352-9. doi: 10.1200/JCO.2012.44.1477. Epub 2012 Nov 13. PMID 23150706
- [Result] Kohno T, Ichikawa H, Totoki Y, Yasuda K, Hiramoto M, Nammo T, Sakamoto H, Tsuta K, Furuta K, Shimada Y, Iwakawa R, Ogiwara H, Oike T, Enari M, Schetter AJ, Okayama H, Haugen A, Skaug V, Chiku S, Yamanaka I, Arai Y, Watanabe S, Sekine I, Ogawa S, Harris CC, Tsuda H, Yoshida T, Yokota J, Shibata T. KIF5B-RET fusions in lung adenocarcinoma. Nat Med. 2012 Feb 12;18(3):375-7. doi: 10.1038/nm.2644. PMID 22327624
- [Result] Lipson D, Capelletti M, Yelensky R, Otto G, Parker A, Jarosz M, Curran JA, Balasubramanian S, Bloom T, Brennan KW, Donahue A, Downing SR, Frampton GM, Garcia L, Juhn F, Mitchell KC, White E, White J, Zwirko Z, Peretz T, Nechushtan H, Soussan-Gutman L, Kim J, Sasaki H, Kim HR, Park SI, Ercan D, Sheehan CE, Ross JS, Cronin MT, Janne PA, Stephens PJ. Identification of new ALK and RET gene fusions from colorectal and lung cancer biopsies. Nat Med. 2012 Feb 12;18(3):382-4. doi: 10.1038/nm.2673. PMID 22327622
- [Result] Takeuchi K, Soda M, Togashi Y, Suzuki R, Sakata S, Hatano S, Asaka R, Hamanaka W, Ninomiya H, Uehara H, Lim Choi Y, Satoh Y, Okumura S, Nakagawa K, Mano H, Ishikawa Y. RET, ROS1 and ALK fusions in lung cancer. Nat Med. 2012 Feb 12;18(3):378-81. doi: 10.1038/nm.2658. PMID 22327623
- [Result] Plaza-Menacho I, Mologni L, McDonald NQ. Mechanisms of RET signaling in cancer: current and future implications for targeted therapy. Cell Signal. 2014 Aug;26(8):1743-52. doi: 10.1016/j.cellsig.2014.03.032. Epub 2014 Apr 3. PMID 24705026
- [Result] Drilon A, Wang L, Hasanovic A, Suehara Y, Lipson D, Stephens P, Ross J, Miller V, Ginsberg M, Zakowski MF, Kris MG, Ladanyi M, Rizvi N. Response to Cabozantinib in patients with RET fusion-positive lung adenocarcinomas. Cancer Discov. 2013 Jun;3(6):630-5. doi: 10.1158/2159-8290.CD-13-0035. Epub 2013 Mar 26. PMID 23533264
- [Result] Michels S, Scheel AH, Scheffler M, Schultheis AM, Gautschi O, Aebersold F, Diebold J, Pall G, Rothschild S, Bubendorf L, Hartmann W, Heukamp L, Schildhaus HU, Fassunke J, Ihle MA, Kunstlinger H, Heydt C, Fischer R, Nogova L, Mattonet C, Hein R, Adams A, Gerigk U, Schulte W, Luders H, Grohe C, Graeven U, Muller-Naendrup C, Draube A, Kambartel KO, Kruger S, Schulze-Olden S, Serke M, Engel-Riedel W, Kaminsky B, Randerath W, Merkelbach-Bruse S, Buttner R, Wolf J. Clinicopathological Characteristics of RET Rearranged Lung Cancer in European Patients. J Thorac Oncol. 2016 Jan;11(1):122-7. doi: 10.1016/j.jtho.2015.09.016. PMID 26762747
- [Result] Gautschi O, Zander T, Keller FA, Strobel K, Hirschmann A, Aebi S, Diebold J. A patient with lung adenocarcinoma and RET fusion treated with vandetanib. J Thorac Oncol. 2013 May;8(5):e43-4. doi: 10.1097/JTO.0b013e31828a4d07. No abstract available. PMID 23584301
- [Result] Kodama T, Tsukaguchi T, Satoh Y, Yoshida M, Watanabe Y, Kondoh O, Sakamoto H. Alectinib shows potent antitumor activity against RET-rearranged non-small cell lung cancer. Mol Cancer Ther. 2014 Dec;13(12):2910-8. doi: 10.1158/1535-7163.MCT-14-0274. Epub 2014 Oct 27. PMID 25349307
- [Result] Choueiri TK, Escudier B, Powles T, Mainwaring PN, Rini BI, Donskov F, Hammers H, Hutson TE, Lee JL, Peltola K, Roth BJ, Bjarnason GA, Geczi L, Keam B, Maroto P, Heng DY, Schmidinger M, Kantoff PW, Borgman-Hagey A, Hessel C, Scheffold C, Schwab GM, Tannir NM, Motzer RJ; METEOR Investigators. Cabozantinib versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1814-23. doi: 10.1056/NEJMoa1510016. Epub 2015 Sep 25. PMID 26406150
- [Result] Choueiri TK, Escudier B, Powles T, Tannir NM, Mainwaring PN, Rini BI, Hammers HJ, Donskov F, Roth BJ, Peltola K, Lee JL, Heng DYC, Schmidinger M, Agarwal N, Sternberg CN, McDermott DF, Aftab DT, Hessel C, Scheffold C, Schwab G, Hutson TE, Pal S, Motzer RJ; METEOR investigators. Cabozantinib versus everolimus in advanced renal cell carcinoma (METEOR): final results from a randomised, open-label, phase 3 trial. Lancet Oncol. 2016 Jul;17(7):917-927. doi: 10.1016/S1470-2045(16)30107-3. Epub 2016 Jun 5. PMID 27279544
- [Result] Choueiri TK, Halabi S, Sanford BL, Hahn O, Michaelson MD, Walsh MK, Feldman DR, Olencki T, Picus J, Small EJ, Dakhil S, George DJ, Morris MJ. Cabozantinib Versus Sunitinib As Initial Targeted Therapy for Patients With Metastatic Renal Cell Carcinoma of Poor or Intermediate Risk: The Alliance A031203 CABOSUN Trial. J Clin Oncol. 2017 Feb 20;35(6):591-597. doi: 10.1200/JCO.2016.70.7398. Epub 2016 Nov 14. PMID 28199818
- [Result] Kurzrock R, Sherman SI, Ball DW, Forastiere AA, Cohen RB, Mehra R, Pfister DG, Cohen EE, Janisch L, Nauling F, Hong DS, Ng CS, Ye L, Gagel RF, Frye J, Muller T, Ratain MJ, Salgia R. Activity of XL184 (Cabozantinib), an oral tyrosine kinase inhibitor, in patients with medullary thyroid cancer. J Clin Oncol. 2011 Jul 1;29(19):2660-6. doi: 10.1200/JCO.2010.32.4145. Epub 2011 May 23. PMID 21606412
- [Result] Vergote IB, Smith DC, Berger R, Kurzrock R, Vogelzang NJ, Sella A, Wheler J, Lee Y, Foster PG, Weitzman R, Buckanovich RJ. A phase 2 randomised discontinuation trial of cabozantinib in patients with ovarian carcinoma. Eur J Cancer. 2017 Sep;83:229-236. doi: 10.1016/j.ejca.2017.06.018. Epub 2017 Jul 26. PMID 28755607
- [Result] Mukhopadhyay S, Pennell NA, Ali SM, Ross JS, Ma PC, Velcheti V. RET-rearranged lung adenocarcinomas with lymphangitic spread, psammoma bodies, and clinical responses to cabozantinib. J Thorac Oncol. 2014 Nov;9(11):1714-9. doi: 10.1097/JTO.0000000000000323. PMID 25436805
- [Result] Drilon A, Rekhtman N, Arcila M, Wang L, Ni A, Albano M, Van Voorthuysen M, Somwar R, Smith RS, Montecalvo J, Plodkowski A, Ginsberg MS, Riely GJ, Rudin CM, Ladanyi M, Kris MG. Cabozantinib in patients with advanced RET-rearranged non-small-cell lung cancer: an open-label, single-centre, phase 2, single-arm trial. Lancet Oncol. 2016 Dec;17(12):1653-1660. doi: 10.1016/S1470-2045(16)30562-9. Epub 2016 Nov 4. PMID 27825636